CLINICAL TRIAL: NCT05242445
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Single Doses of Cetrelimab (JNJ 63723283), an Anti-PD-1 Monoclonal Antibody, in Virologically Suppressed Participants With Chronic Hepatitis B Virus Infection
Brief Title: A Study of Cetrelimab in Participants With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CR109158; 2021-004857-21 (EudraCT Number); 63723283HPB1001 (Other: Janssen Research and Development, LLC)
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: Cetrelimab or Placebo (Dose 1) (Experimental): Participants will receive cetrelimab Dose 1 or placebo via subcutaneous (SC) injection on Day 1.
  Interventions: Drug: Cetrelimab; Drug: Placebo
- Cohort 2 (Optional): Cetrelimab or Placebo (Dose 2) (Experimental): Participants will receive cetrelimab Dose 2 or placebo administered via an Intravenous (IV) infusion on Day 1 based on the data review of previous cohort(s) (safety and tolerability data through at least 6 weeks postdose as well as pharmacokinetic (PK) and receptor occupancy (RO) data through at least day 4 postdose).
  Interventions: Drug: Cetrelimab; Drug: Placebo
- Cohort 3 (Optional): Cetrelimab or Placebo (Experimental): Participant will receive cetrelimab or placebo via SC injection based on the data review of previous cohort(s) (safety and tolerability data through at least 6 weeks postdose as well as PK and RO data through at least day 4 postdose).
  Interventions: Drug: Cetrelimab; Drug: Placebo
- Cohort 4 (Optional): Cetrelimab or Placebo (Experimental): Participant will receive cetrelimab or placebo via SC injection based on the data review of previous cohorts (safety and tolerability data through at least 6 weeks postdose as well as PK and RO data through at least day 4 postdose).
  Interventions: Drug: Cetrelimab; Drug: Placebo

INTERVENTIONS:
Drug: Cetrelimab — Cetrelimab (Dose 1 and Dose 2) will be administered via SC injection or as an IV infusion.
  Other Names: JNJ-63723283
Drug: Placebo — Placebo will be administered via SC injection or as an IV infusion.

SUMMARY:
The purpose of the study is to characterize the pharmacokinetic (PK) profile of cetrelimab administered subcutaneous (SC) and optionally intravenous (IV) in chronic hepatitis B (CHB) participants.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a small deoxyribonucleic acid (DNA) virus that infects the liver and can cause either acute (less than 6 months) or chronic (more than 6 months) infection. Persistence of HBV infection requires antigen-specific immune tolerance that prevents clearance of infected cells. Cetrelimab (JNJ-63723283) is a fully human immunoglobulin (Ig) G4 kappa monoclonal antibody (mAb) that binds to programmed cell death receptor-1 (PD-1) with high affinity and specificity. PD-(L)1 inhibitors could possibly reverse the immune dysfunction from HBV. The study will be conducted in 3 phases: a screening phase (6 weeks), a single dose intervention phase (1 day), and a 24-week follow-up phase. The duration of individual participation will be up to 30 weeks. Key safety assessments include monitoring of Adverse Events (AEs), physical examination, vital signs, Electrocardiogram (ECGs), Injection site reaction (ISRs), Infusion-related reaction (IRRs), and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Must have chronic hepatitis B virus (HBV) infection documented
* Participants should be virologically suppressed, Hepatitis Be antigen (HBeAg) status (positive or negative) be on stable Nucleotide analog (NA) treatment for at least 6 months
* Must have: a) A liver biopsy result classified as Metavir F0-F2 within 2 years prior to screening; b) If a liver biopsy result is not available: Fibroscan liver stiffness measurement less than or equal to (<=) to 9.0 kilopascals (kPa) within 6 months prior to screening or at the time of screening
* Must be medically stable
* Must have a body mass index (weight in kilogram [kg] divided by the square of height in meters) between 18.0 and 30.0 kilograms per meter square (kg/m^2), extremes included

Exclusion Criteria

* History or evidence of clinical signs or symptoms of hepatic decompensation, including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices
* Participants with evidence of liver disease of non-HBV etiology.
* Participants with history or signs of cirrhosis or portal hypertension (nodules, no smooth liver contour, no normal portal vein, spleen size greater than or equal to [>=] 12 centimeters) or signs of hepatocellular carcinoma (HCC) on an abdominal ultrasound performed within 6 months prior to screening or at the time of screening
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Cetrelimab | Up to 24 weeks
  Cmax is defined as maximum observed serum concentration of cetrelimab.
Area Under the Concentration-time Curve From Time Zero to Last Measurable Concentration (AUC[0-last]) of Cetrelimab | Up to 24 weeks
  AUC(0-last) is defined as area under the concentration-time curve from time 0 to the time of the last measurable concentration (non-below quantification limit [non-BQL]) of cetrelimab as calculated by linear-linear trapezoidal summation.
Apparent Terminal Elimination Half-life (t1/2) of Cetrelimab | Up to 24 weeks
  t1/2 is defined as apparent terminal elimination half-life of cetrelimab.
Total Systemic Clearance of Cetrelimab | Up to 24 weeks
  Total systemic clearance is a quantitative measure of the rate at which cetrelimab is removed from the body.

SECONDARY OUTCOMES:
Change from Baseline in HBsAg and HBeAg Levels Over Time | Baseline up to 30 weeks
  Change from baseline in Hepatitis B surface antigen (HBsAg), Hepatitis Be antigen (HBeAg) levels over time will be reported.
Change from Baseline in Hepatitis B Virus Deoxyribonucleic acid (HBV DNA) Levels Over Time | Baseline up to 30 weeks
  Change from baseline in HBV DNA levels over time will be reported.
Number of Participants with Adverse Events (AEs) | Up to 30 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Cohorts 1,3 and 4: Number of Participants with Injection Site Reaction (ISR) | Up to 30 weeks
  Number of Participants with ISR will be reported. An ISR is any adverse reaction at a subcutaneous (SC) study intervention injection-site.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 30 weeks
  Number of participants with abnormalities in clinical laboratory tests (including hematology, serum chemistry and urinalysis) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (13):
- Belgium (2):
  - SGS Belgium NV, Edegem
  - Az Sint-Maarten, Mechelen
- France (4):
  - Hopital Beaujon, Clichy
  - APHP - Hopital Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - Hopital Saint-Antoine, Paris
- Germany (2):
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
- Poland (2):
  - PUNKT ZDROWIA Hlebowicz Jakubowski Lekarze sp.p., Gdansk
  - ID Clinic, Mysłowice
- Spain (3):
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Gral. Univ. Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency